CLINICAL TRIAL: NCT04743271
Title: Uncovering the Impact of Diet on the Human Circadian Timing System
Brief Title: Food and Circadian Timing
Acronym: FACT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Andrew McHill, Principal Investigator, Oregon Health and Science University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: STUDY00022478
Record Dates: First submitted 2021-01-28; First posted 2021-02-08 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Diet, High-Fat; Circadian Rhythm
Keywords: Circadian Rhythm; High Fat; Diet
MeSH Terms: interventions — Diet, High-Fat; Diet, Fat-Restricted

STUDY DESIGN:
Masking Description: As it will be easy to discern meal fat content, participant blinding is not possible. Participants will be blinded to clock time and light-dark cues and statisticians will be blinded of condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-Fat Diet (Experimental): 50% fat, 35% carbohydrate and 15% protein; 33% of each mono, poly and saturated fat
  Interventions: Other: High-Fat Diet
- Low-Fat Diet (Active Comparator): 30% fat, 55% carbohydrate and 15% protein
  Interventions: Other: Low-Fat Diet

INTERVENTIONS:
Other: High-Fat Diet — The diet will consist of a breakfast, lunch, dinner, and snack
  Arms: High-Fat Diet
Other: Low-Fat Diet — The diet will consist of a breakfast, lunch, dinner, and snack
  Arms: Low-Fat Diet

SUMMARY:
The goals of this study are to uncover the influence of diet on the human circadian timing system. The protocol is a 46-day (28 outpatient days, 18 inpatient days over two 9 day visits) randomized cross-over study designed to elucidate the speed of entrainment in response to a high-fat diet.

DETAILED DESCRIPTION:
Synchronization of the timing of biological processes and behaviors with the 24-hour light-dark cycle is fundamental to almost every physiological process, cognitive function, and overall health. As the average circadian period in humans is ~9 min longer than the 24-h day, and artificial lighting allows a further delay in the clock, circadian entrainment must occur every day. This makes the process of circadian entrainment of the internal clock with the external environment a commonly overlooked process, but one that has serious ramifications if impaired.

In rodent models, high-fat diets have been shown to disorganize the circadian timing system. There has been limited examination, however, of how composition of diet acts on the circadian timing system in humans. The ability to entrain to a new light schedule has been briefly examined after a high-fat diet in rodent models.When mice are exposed to a 6-h shift in the light-dark cycle and fed a diet composed of ~50% fat for 3 weeks, they experience a 20% slower rate of re-entrainment to the new light cycle as compared to mice fed a low-fat diet. Further, these mice had an attenuated response to a phase-advancing light pulse. Moreover, simply providing a high-fat diet to mice results in a lengthened circadian period and a shift in ad libitum eating patterns into the typical rest phase.

The goals of this study are to uncover the influence of diet on the human circadian timing system. The protocol is a 46-day (28 outpatient days, 18 inpatient days over two 9 day visits) randomized cross-over study designed to elucidate the speed of entrainment in response to a high-fat diet. Participants will be provided 3 weeks of a high-fat diet (2-weeks outpatient, 1-week inpatient) of 50% calories from fat. The protocol includes two types of data collection; ambulatory monitoring on strict sleep-wake schedules with either high-fat or low-fat meals provided by the study team and precise in-laboratory measurements of circadian timing, entrainment, and other physiological markers of sleep and cardiometabolic health.

1. Ambulatory Monitoring: Participants will maintain a consistent 14-day at home 8h sleep schedule at habitual times before both laboratory visits to ensure 1) subjects are not sleep restricted and 2) that they are obtaining the same light-dark schedule prior to each laboratory visit for stable entrainment; verified by actigraphy, sleep logs, and call-ins to a time stamped recorder. Drugs, medications, caffeine, alcohol, and nicotine will be proscribed during this time and toxicology analysis will be performed upon in-laboratory admission.
2. Outpatient diet: For 2-weeks prior to each protocol, participants will consume an outpatient isocaloric diet designed to meet individual daily energy requirements; diet designed and prepared by investigators. Diets will either be designed to be high in calories from fat (50% fat, 35% carbohydrate and 15% protein; 33% of each mono, poly and saturated fat) or low-fat (30% fat, 55% carbohydrate and 15% protein) (randomized-crossover design). The diet will consist of a breakfast, lunch, dinner, and snack and participants will either come to the laboratory ~3 days or staff will deliver meals. Participants will be instructed to only consume the food provided during these 14-days. Adherence to the diet will be captured via tracking meals using a mobile food tracking application (MealLogger AppTM (Wellness Foundry, New York)).
3. Inpatient Protocols: Participants will be admitted to an individual room free of external time cues (e.g., clocks, radios, computers, visitors and sunlight). Room temperature is maintained at 21 - 22.2 °C and light intensity set at ≤5 lux during scheduled constant posture procedures, room light (400 lux) during entrainment wakefulness and 0 lux (darkness) during scheduled sleep opportunities. Participants will be instrumented for full polysomnography (PSG), electrocardiogram, and a rectal thermistor for continuous core body temperature measurement. An 18-gauge IV catheter will also be inserted into the forearm and connected to a triple-stopcock manifold via an IV loop with a 12- foot small-lumen extension cable through which blood sampling can continue in the next room without disturbing sleep.

After instrumentation, participants will be given a sleep opportunity and will awakened to dim-lighting and maintaining a constant posture protocol for accurate assessment of circadian phase, resting metabolic rate, and other physiological outcomes. After the constant posture protocol, participants' light-dark cycle will be changed for 6 identical days, followed by a second constant posture protocol for re-assessment of circadian phase. This protocol will be repeated while participants are provided the other cross-over meal. Investigators/nurses will be present in the lab or in a central control room 24 h per day to monitor subject health, data acquisition, provide meals, collect biologic specimens, perform tests, and record sleep. A physician is always on call when a participant is in the laboratory. An extensive series of protocols and checklists and team practices are used to ensure uniformity in execution of standard procedures.

Energy content of diets will be designed to meet individual daily energy requirements. Dietitians will prepare isocaloric meals containing macronutrient contents of high or low-fat diet and no caffeine. Caloric intake will be the same caloric and macronutrient composition for each day of laboratory study and will be provided as miniature snacks frequently during each constant posture protocol (e.g., ¼ turkey & cheese sandwich, juice and water).

ELIGIBILITY:
Inclusion Criteria:

* Healthy, lean men and women

Exclusion Criteria:

* Major dietary restrictions (such as entirely dairy-free and/or meat-free diets)
* A body mass index (BMI) of 18.5< [BMI] < 24.9 kg/m^2 and a waist circumference <94/80cm
* Currently psychiatrically/psychologically unsuitable for participation
* Drug/alcohol use, including smoking
* Medication/drug use, including prescribed and over-the-counter medications
* History of working irregular day and night hours, regular night work, or rotating shift work for the 1 year prior to the study.
* Traveled across more than 1 time zone during the 3 months prior to the study
* Currently consuming a habitual high-fat diet
* Chronobiologic and sleep disorders
* Diseases of the Cardiovascular System
* Metabolic Syndrome; Two or more of these factors will be excluded from the study:

  1. HDL cholesterol of less than 40 mg/dL in men or less than 50 mg/dL in women;
  2. systolic blood pressure>135 mmHg or diastolic blood pressure>85 mmHg;
  3. Fasting blood glucose ≥ 100 mg/dL;
  4. Triglycerides ≥ 150 mg/dL.
* Pre-Diabetes/Diabetes
* Hypertension
* Disorders of the Respiratory System
* Disorders of the Kidney and Urinary Tract
* Infectious Diseases
* Disorders of the Gastrointestinal System
* Disorders of the Immune System
* Disorders of the Hematopoietic System
* Neoplastic Diseases
* Endocrine and Metabolic Diseases
* Neurologic Disorders
* Subjects must not be currently participating in another research study that would influence their safe participation in our study

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in Speed of entrainment | Over 18 days
  Entrainment will be determined as a stable phase angle between sleep and both melatonin onset. Blood and/or saliva will be assayed for melatonin using standardized assays. Melatonin onset will be calculated using the linear interpolated time at which melatonin levels reach 25% of a fitted peak-to-trough amplitude. This will be analyzed using phase angle between sleep and melatonin onset.

SECONDARY OUTCOMES:
Change in Phase Angle of entrainment | Over 18 days
  Phase angle will be calculated as dim-light melatonin onset minus sleep onset during each constant posture protocol. Differences in phase angle of entrainment between sleep and melatonin onset will be first examined using planned comparison dependent t-tests between the high-fat and low-fat visits. The study will use planned comparison dependent t-tests to compare phase angle of entrainment from constant posture day 1 vs constant posture day 2 to uncover potential differences in phase angle in response to an advance in light exposure under differing diet conditions
Change in Core Body Temperature Entrainment | Over 18 days
  Core body temperature entrainment will be determined as a stable phase angle between sleep and core body temperature minimum. Temperature data will be collected every minute though rectal thermistors.
Change in Core Body Temperature Phase angle of Entrainment | Over 18 days
  Core body temperature entrainment will be determined as core body temperature minimum minus sleep onset. Temperature data will be collected every minute though rectal thermistors.
Change in glucose tolerance | Over 18 days
  The participant's glucose and insulin response to a mixed meal diet high in carbohydrates may be tested. During this mixed meal test, a baseline blood draw will occur ~7-min before the meal and then the frequency of blood samples will increase to every 10-min after the meal for 90 min and then every 30 min for 90 min for a total of 12 samples over 180 min to measure glucose and hormone response in detail. Examined using planned comparison dependent t-tests between the high-fat and low-fat visits.
Change in Energy Metabolism | Over 18 days
  Resting energy metabolism will be measured every ~4h via indirect calorimetry. Examined using planned comparison dependent t-tests between the high-fat and low-fat visits.
Change in Blood Pressure | Over 18 days
  Resting blood pressure will be measured every ~2h via blood pressure cuff. Examined using planned comparison dependent t-tests between the high-fat and low-fat visits.
Change in Heart Rate | Over 18 days
  Resting heart rate will be measured every ~2h via blood pressure cuff. Examined using planned comparison dependent t-tests between the high-fat and low-fat visits.
Change in Malondialdehyde | Over 18 days
  Malondialdehyde will be measured every ~4h via blood from IV catheter. Examined using planned comparison dependent t-tests between the high-fat and low-fat visits.
Change in Total Antioxidant Capacity | Over 18 days
  Total Antioxidant Capacity will be measured every ~4h via blood from IV catheter. Examined using planned comparison dependent t-tests between the high-fat and low-fat visits.
Change in C-reactive protein | Over 18 days
  C-reactive protein will be measured every ~4h via blood from IV catheter. Examined using planned comparison dependent t-tests between the high-fat and low-fat visits.
Change in TNF-alpha | Over 18 days
  TNF-alpha will be measured every ~4h via blood from IV catheter. Examined using planned comparison dependent t-tests between the high-fat and low-fat visits.
Change in Triglycerides | Over 18 days
  Triglycerides will be measured every ~4h via blood from IV catheter. Examined using planned comparison dependent t-tests between the high-fat and low-fat visits.
Change in Fatty Acids | Over 18 days
  Fatty acids will be measured every glucose tolerance test from IV catheter. Examined using planned comparison dependent t-tests between the high-fat and low-fat visits.
Change in Vascular Endothelial Function | Over 18 days
  We will measure vascular endothelial function starting ~10-min after each awakening in a constant posture following a fast. Brachial artery flow-mediated dilation will be measured in the supine position. Examined using planned comparison dependent t-tests between the high-fat and low-fat visits.
Change in Psychomotor Vigilance Task | Over 18 days
  The psychomotor vigilance task will be administered via computer test every 2h to assess sustained attention. Examined using planned comparison dependent t-tests between the high-fat and low-fat visits.
Change in Digit Symbol Substitution Task | Over 18 days
  The digit symbol substitution task will be administered via computer test every 2h to assess attention and accuracy. Examined using planned comparison dependent t-tests between the high-fat and low-fat visits.
Change in Addition Task | Over 18 days
  The addition task will be administered via computer test every 2h to assess working memory. Examined using planned comparison dependent t-tests between the high-fat and low-fat visits.
Change in Subjective Alertness | Over 18 days
  Visual analog scales will be administered via computer test every 2h to subjective alertness. Examined using planned comparison dependent t-tests between the high-fat and low-fat visits.
Change in Profile of Mood States | Over 18 days
  Profile of mood states (POMS scale) will be administered via paper questionnaire every 2h to subjective alertness. Examined using planned comparison dependent t-tests between the high-fat and low-fat visits.
Change in Positive and Negative Affect Schedule | Over 18 days
  Positive and negative affect schedule (PANAS scale) will be administered via paper questionnaire every 2h to subjective alertness. Examined using planned comparison dependent t-tests between the high-fat and low-fat visits.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew McHill, PhD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No